CLINICAL TRIAL: NCT04827888
Title: The Effect Of BMI On Thirty-day Postoperative Morbidities And Mortality For The Most Common Orthopaedic Procedures
Brief Title: Effect of BMI on Postoperative Morbidities of Orthopaedic Procedures
Acronym: BMIORTHO
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Muhyeddine Al-Taki, Assistant Professor of Clinical Surgery, American University of Beirut Medical Center
Other Study IDs: 20210330BMI
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Orthopedic Procedures; Obesity
Keywords: weight; orthopedic surgery; BMI; Post-Op Complication
MeSH Terms: conditions — Obesity; Body Weight; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- underweight: patients who underwent one of the 25 common orthopaedic surgeries and have a body mass index (BMI) of <18.5kg/m2
  Interventions: Procedure: Orthopaedic surgery
- normal-weight: patients who underwent one of the 25 common orthopaedic surgeries and have a BMI between 18.5kg/m2 and 24.9kg/m2
  Interventions: Procedure: Orthopaedic surgery
- overweight: patients who underwent one of the 25 common orthopaedic surgeries and have a BMI between 25kg/m2 and 29.9kg/m2
  Interventions: Procedure: Orthopaedic surgery
- mildly obese: patients who underwent one of the 25 common orthopaedic surgeries and have a BMI between 30kg/m2 and 34.9kg/m2
  Interventions: Procedure: Orthopaedic surgery
- moderately-to-severely obese: patients who underwent one of the 25 common orthopaedic surgeries and have a BMI ≥35kg/m2
  Interventions: Procedure: Orthopaedic surgery

INTERVENTIONS:
Procedure: Orthopaedic surgery — One of the 25 most common orthopedic surgeries reported in the database which are the following as per surgical types: spine surgery (CPT codes 63030, 63047, 22612, 22551 or 22558), trauma (CPT codes 27236, 27125, 27244, 27814, or 27792), sports medicine injuries (CPT codes 29881, 29827, 29880, 29888, 29826, 29877, 29807, or 23412), or joint arthroplasty (CPT codes 27447, 27130, 23472, 27487, 27134, 27446, or 27486).

SUMMARY:
Obesity is associated with poor surgical outcome and complications. The literature does not provide a comprehensive view on the effect of body mass index (BMI) on perioperative outcomes in orthopedic surgeries. Therefore, we aim to determine the effect of BMI on 30-day perioperative outcomes in patients undergoing the first 25 most commonly performed orthopedic surgeries using a retrospective cohort study design. The knowledge of the effect of BMI on orthopedic surgeries will improve the knowledge of surgeons about the expected morbidities.

DETAILED DESCRIPTION:
Obesity is associated with poor surgical outcome and complications. The literature does not provide a comprehensive view on the effect of body mass index (BMI) on perioperative outcomes in orthopedic surgeries. Therefore, we aim to determine the procedure specific, independent-effect of BMI on 30-day perioperative outcomes in patients undergoing the first 25 most commonly performed orthopedic surgeries.

The study is a retrospective cohort study. The subjects will be the individuals undergoing one of first 25 most commonly performed orthopedic surgeries, whose information is derived form the de-identified patients' data collected through the American College of Surgeons National Surgical Quality Improvement Program (ACS-NSQIP) database. The primary outcome will be composite post-operative morbidity. Specific morbidities will also be evaluated including cardiovascular, vascular and renal complications, length-of-stay (LOS), and the need for re-intervention and readmission, as well as 30-day mortality. Descriptive statistics and multivariable regression models will assess the independent-effect of BMI on outcomes.

The knowledge of the effect of BMI on orthopedic surgeries will improve the knowledge of surgeons about the expected morbidities. The surgeon will be able to better counsel obese patients and devise a better surgical plan to prevent or deal with the expected outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion and exclusion criteria are the same as that of ACS-NSQIP database.
* All patients who have undergone any of the 25 most common orthopedic procedures as primary procedure as identified through the CPT codes

Exclusion Criteria:

* All patients whose BMI was not reported

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Representative of the population from ACS-NSQIP
Sampling Method: Non-Probability Sample
Enrollment: 76189 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Composite morbidity | within the 30 days following the surgery
  Composite morbidity is defined as the presence of any of the specific morbidities during the 30-days following surgery as recorded in the ACS-NSQIP database. The odds ratio of composite morbidity for each BMI group will be calculated as compared to normal-weight group.

SECONDARY OUTCOMES:
mortality | within the 30 days following the surgery
  odds ratio of mortality within the 30-days following the surgery for each BMI group as compared to normal-weight group
wound | within the 30 days following the surgery
  odds ratio of specific morbidity of surgical wound for each BMI group as compared to normal-weight group
cardiac | within the 30 days following the surgery
  specific morbidity of cardiac complication for each BMI group as compared to normal-weight group
respiratory | within the 30 days following the surgery
  odds ratio of specific morbidity of respiratory complication
urinary | within the 30 days following the surgery
  odds ratio of specific morbidity of urinary complication for each BMI group as compared to normal-weight group
neurological | within the 30 days following the surgery
  odds ratio of specific morbidity of neurological (CNS) complication for each BMI group as compared to normal-weight group
thromboembolism | within the 30 days following the surgery
  odds ratio of specific morbidity of thromboembolism for each BMI group as compared to normal-weight group
sepsis | within the 30 days following the surgery
  odds ratio of specific morbidity of sepsis for each BMI group as compared to normal-weight group
bleeding | within the 30 days following the surgery
  odds ratio of bleeding or transfusion need for each BMI group as compared to normal-weight group
Re-op | within the 30 days following the surgery
  odds ratio of need for re-admission/re-operation for each BMI group as compared to normal-weight group

CONTACTS AND LOCATIONS:
Overall Officials: Muhyeddine Al-Taki, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
Only the de-identified and coded data are available through the registry and we do not plan of sharing any individual data